CLINICAL TRIAL: NCT04500509
Title: Diclofenac Potassium With or Without Vaginal Dinoprostone Prior to Hysterosalpingography in Primarily Infertile Patients: a Randomized Controlled Trial
Brief Title: Diclofenac Potassium With or Without Vaginal Dinoprostone Prior to Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/352/3/19
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Diclofenac; Dinoprostone

STUDY DESIGN:
Intervention Model Description: double blind placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind placebo controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): patients will have of oral diclofenac potassium 60 minutes before the procedure plus one tablets of vaginal dinoprostone (6 mg) 6 hours prior to the procedure
  Interventions: Drug: diclofenac potassium + dinoprostone
- Group B (Placebo Comparator): patients will have of oral diclofenac potassium 60 minutes before the procedure plus one tablets of vaginal placebo 6 hours prior to the procedure
  Interventions: Drug: diclofenac potassium + placebo

INTERVENTIONS:
Drug: diclofenac potassium + dinoprostone — patients will have of oral diclofenac potassium 60 minutes before the procedure plus one tablets of vaginal dinoprostone (6 mg) 6 hours prior to the procedure by the patient
  Arms: Group A
Drug: diclofenac potassium + placebo — patients will have of oral diclofenac potassium 60 minutes before the procedure plus one tablets of vaginal placebo 6 hours prior to the procedure by the patient
  Arms: Group B

SUMMARY:
The aim of our study is to determine the efficacy of oral diclofenac potassium with or without vaginal dinoprostone prior to hysterosalpingography in primarily infertile patients on the pain scores during HSG.

DETAILED DESCRIPTION:
hysterosalpingography is a diagnosis procedure in the evaluation of infertile women and considered to be the traditional and the gold standard in the assessment of the patency of the fallopian tubes. The major disadvantage of hysterosalpingography is pain. In a study reported the patients complained of moderate to severe pain during the procedure. It is reported that some patients undergoing hysterosalpingography was more stressful and anxiety and effect on pain scores.

ELIGIBILITY:
Inclusion Criteria:

* primary infertility female came for HSG

Exclusion Criteria:

* any patient has contraindication to HSG

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — primary infertility female
Enrollment: 200 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Mean pain score during hysterosalpigography by visual analog scale | 15 minutes
  pain during hysterosalpigography assessed by the visual analog scale from 0=no pain to 10 = the worst pain imaginable

SECONDARY OUTCOMES:
Intensity of pain | 30 minutes after the procedure
  Pain intensity will be assessed by visual analogue scale 30 minutes after the procedure.visual analogue scale ranging from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No